CLINICAL TRIAL: NCT07262359
Title: A Multi-Center, Prospective, Observational Registry for the Evaluation of Coronary Artery Calcified Nodules Using Intravascular Ultrasound (IVUS) and/or Optical Coherence Tomography (OCT) in China (CN-IVI Registry)
Brief Title: Intravascular Imaging Evaluated Calcified Nodule China Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The First Hospital of Jilin University (Other); Zhongnan Hospital (Other); Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Sponsor
Other Study IDs: CN-IVI Registry
Record Dates: First submitted 2025-09-29; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Coronary Artery Atherosclerosis; Coronary Calcified Nodules; Coronary Calcification
Keywords: coronary artery disease; coronary calcification; coronary calcified nodules; optical coherence tomography; intravascular ultrosound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is this study about? This is a nationwide research study in China focused on understanding a specific type of challenging plaque in heart arteries called a Calcified Nodule (CN). The study will use advanced imaging technology inside the blood vessels to see these nodules in great detail, track how they are treated, and see how patients do in the long term.

Why is this important? Calcified nodules are hard, bony-like plaques that can cause sudden heart attacks. They are difficult to treat with standard procedures like stenting because they are rigid and can be unpredictable. This registry aims to create a large database of real-world cases to help doctors better understand how to identify and manage CNs effectively, ultimately improving patient care and outcomes across China.

What are IVUS and OCT? These are sophisticated imaging tools that doctors use during a heart catheterization. Think of them like a "GPS" or an "ultrasound" for the inside of your arteries.

IVUS (Intravascular Ultrasound): Uses sound waves to create a detailed, 360-degree picture of the artery wall. It shows the size of the plaque and how deep it goes, helping doctors choose the right size stent.

OCT (Optical Coherence Tomography): Uses light waves to create extremely high-resolution images, like a microscope inside the artery. It is excellent for seeing the precise surface and structure of a calcified nodule.

Together, these tools give doctors a clear view of the problem, which is crucial for planning the best treatment strategy.

What will the study do?

The registry will collect anonymous data from participating hospitals across China. Researchers will analyze:

How common calcified nodules are in Chinese patients.

The best ways to use IVUS and OCT to identify and characterize CNs.

Which treatment techniques (e.g., special balloons, atherectomy) work best.

The long-term results for patients who receive stents to treat a CN.

Who is this for?

Patients & Families: To understand that advanced care and research are being dedicated to complex heart conditions. Participation (if eligible) contributes to medical knowledge that may help future patients.

Healthcare Providers: To provide a standardized, large-scale analysis of CNs, leading to improved diagnosis, treatment guidelines, and procedural techniques for this complex lesion.

This registry represents a significant step forward in personalized cardiac care in China, using cutting-edge technology to solve a difficult clinical problem.

DETAILED DESCRIPTION:
1. Study Title and Overview

   Official Title: A Multi-Center, Prospective, Observational Registry for the Evaluation of Coronary Artery Calcified Nodules Using Intravascular Ultrasound (IVUS) and/or Optical Coherence Tomography (OCT) in China (CN-IVI Registry)

   Overview: The CN-IVI Registry is a large-scale, observational study conducted across multiple leading cardiac centers in China. Its primary purpose is to systematically investigate a specific, complex, and high-risk type of coronary plaque known as a Calcified Nodule (CN). By leveraging advanced intracoronary imaging techniques, IVUS and/or OCT, the registry aims to create a robust database to improve the diagnosis, characterization, treatment, and long-term outcomes for patients with this challenging lesion.
2. Background and Rationale: Why Focus on Calcified Nodules?

   Coronary artery disease (CAD) involves the buildup of plaque inside the heart's arteries. While there are several types of plaque, Calcified Nodules are among the most complex and dangerous.

   What is a Calcified Nodule? A CN is a specific type of plaque characterized by a sharp, protruding, and often fractured nodule of calcium that erupts through the artery's inner lining (intima). This creates a irregular, bony surface within the blood vessel that is highly thrombogenic (likely to cause blood clots) and is a known cause of sudden acute coronary syndromes (heart attacks).

   The Clinical Challenge: Treating CNs with percutaneous coronary intervention (PCI) - the procedure to open blocked arteries and place stents - is notoriously difficult. Their hard, irregular nature makes it challenging to fully expand a stent. Incomplete stent expansion, known as "stent underexpansion," is a leading cause of stent failure, including restenosis (re-narrowing) and stent thrombosis (a dangerous blood clot within the stent).

   The Role of Intravascular Imaging: Angiography, the standard X-ray technique used during PCI, is a "shadow" of the artery's interior and often fails to accurately depict the complexity of a CN. This is where IVUS and OCT become critical. They act like a high-definition camera and ultrasound inside the artery, allowing interventional cardiologists to:

   Accurately Identify a calcified nodule versus other types of plaque.

   Characterize its size, shape, and extent of calcium.

   Plan the Procedure by choosing the best techniques to modify the calcium (e.g., with high-pressure balloons, scoring balloons, or rotational atherectomy).

   Optimize the Result by ensuring the stent is fully expanded and well-apposed to the vessel wall after implantation.

   Despite their importance, there is a lack of large-scale, real-world data on the prevalence, optimal management, and outcomes of CNs in the Chinese population. This registry seeks to fill that critical knowledge gap.
3. Primary and Secondary Objectives

   The CN-IVI Registry is designed to answer several key questions:

   Primary Objectives:

   To determine the prevalence and natural distribution of calcified nodules in a large, real-world Chinese cohort of patients undergoing PCI with intravascular imaging guidance.

   To establish the diagnostic criteria and imaging characteristics of CNs using both IVUS and/or OCT, creating a standardized definition for Chinese patients.

   Secondary Objectives:

   To evaluate the immediate procedural success rates of PCI for lesions containing CNs, as assessed by intravascular imaging (e.g., rate of stent underexpansion, acute stent malapposition).

   To assess the impact of different calcium modification techniques (e.g., non-compliant balloons, scoring/cutting balloons, rotational/orbital atherectomy, intravascular lithotripsy) on the final stent result.

   To investigate the long-term clinical outcomes for patients with CNs, including:

   Target Lesion Failure (TLF): A composite of cardiac death, target vessel myocardial infarction, and clinically-driven target lesion revascularization (need for a repeat procedure).

   Rates of stent thrombosis.
4. Study Design and Methodology

   Type: Prospective, multi-center, observational registry.

   Participants: Adult patients (≥18 years) undergoing coronary angiography and PCI for stable coronary artery disease or acute coronary syndromes at participating centers in China, in whom the use of IVUS or OCT is clinically indicated and identifies the presence of a calcified nodule.

   Data Collection: All clinical, procedural, and imaging data will be collected prospectively in a centralized, secure electronic database. This includes:

   Patient demographics and cardiovascular risk factors.

   Angiographic data of the target lesion.

   Raw IVUS and OCT imaging sequences, which will be analyzed in a dedicated core lab by independent experts blinded to patient outcomes to ensure consistency and objectivity.

   Detailed procedural data, including devices used and complications.

   Follow-up: Patients will be followed clinically for up to 3 years after the procedure through outpatient visits and telephone interviews to track their long-term health status and any cardiac-related events.
5. What Participation Means

   For Patients: Participation in this registry does not change your standard medical care. The procedures (angiography, PCI, IVUS/OCT) are all performed based on your clinical need and your doctor's judgment. The registry simply involves allowing researchers to anonymously collect and analyze the data and images from your procedure for the purposes of this study. Your personal information will be kept strictly confidential. Your involvement will help advance medical knowledge and improve care for future patients with similar conditions.

   For Families: This research aims to improve the safety and effectiveness of heart procedures for a particularly tricky problem. By supporting your family member's participation, you are contributing to a national effort to establish best practices that could benefit countless others.

   For Healthcare Providers: This registry will provide invaluable, real-world evidence. It will offer deep insights into the imaging phenotypes of CNs, serve as a benchmark for procedural outcomes, and help generate data-driven guidelines for managing these complex lesions. The core lab analysis will also be an educational resource for the interventional cardiology community.
6. Potential Significance and Impact

   The findings from the CN-IVI Registry are expected to have a direct impact on clinical practice:

   Improved Diagnosis: Establish clear, imaging-based criteria for identifying CNs in Chinese patients.

   Better Treatment Strategies: Provide evidence for which calcium modification techniques are most effective for preparing a nodule for stenting, leading to higher procedural success rates.

   Enhanced Patient Safety: By optimizing stent implantation, the study aims to reduce long-term complications like stent failure and heart attacks, improving overall patient prognosis.

   National Guidelines: The data will inform the development of Chinese and international clinical guidelines on the management of heavily calcified coronary lesions.
7. Ethics and Confidentiality

The study will be conducted in full compliance with the Declaration of Helsinki and Chinese regulatory requirements. The protocol will be approved by the Institutional Review Board (IRB) or Ethics Committee at each participating center. Written informed consent will be obtained from every patient before their data is included in the registry. All patient data will be de-identified to ensure absolute privacy and confidentiality.

In summary, the CN-IVI Registry represents a major collaborative effort to tackle a complex problem in interventional cardiology. By harnessing the power of intravascular imaging, it seeks to translate detailed visual data into tangible improvements in patient care and outcomes across China.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years old.

Intracoronary imaging confirms the presence of at least one calcified nodule lesion.

The patient is willing and able to comply with the study procedures and follow-up until the study concludes.

The subject confirms understanding of the study's risks, benefits, and alternative treatments, and has signed the informed consent form approved by the ethics committee prior to any protocol-related procedures.

Exclusion Criteria:

Contraindication to Procedure: Known contraindication to coronary angiography, PCI, or adjunctive pharmacologic therapy (e.g., aspirin, P2Y12 inhibitors, heparin, contrast media) that cannot be adequately managed with standard medical care.

Life Expectancy: Life expectancy of less than 1 year due to non-cardiac comorbid conditions (e.g., active malignancy, advanced organ failure).

Inability to Follow-Up: Inability or unwillingness to comply with the study protocol or scheduled follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age: ≥ 18 years old. Clinical Presentation: Patient presents with stable coronary artery disease, unstable angina, or an acute coronary syndrome (including NSTEMI and STEMI) and is scheduled to undergo coronary angiography and percutaneous coronary intervention (PCI).
  Intravascular Imaging Indication: The use of intravascular imaging (IVUS or OCT) is clinically indicated and used during the PCI procedure at the discretion of the operating interventional cardiologist. Common clinical indications include:
  Assessment of lesion severity and morphology. Guidance for stent sizing and optimization. Evaluation of complex lesions (e.g., calcified, long, bifurcation lesions).
  Target Lesion Identification: The use of IVUS or OCT must identify the presence of a calcified nodule (CN) in at least one native coronary artery lesion. The CN must be confirmed by the core lab according to standardized definitions:
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 3 years
  including A composite of cardiac death, target vessel myocardial infarction, and clinically-driven target lesion revascularization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Matsumura M, Usui E, Noguchi M, Fujimura T, Fall KN, Zhang Z, Nazif TM, Parikh SA, Rabbani LE, Kirtane AJ, Collins MB, Leon MB, Moses JW, Karmpaliotis D, Ali ZA, Mintz GS, Maehara A. Intravascular Ultrasound-Derived Calcium Score to Predict Stent Expansion in Severely Calcified Lesions. Circ Cardiovasc Interv. 2021 Oct;14(10):e010296. doi: 10.1161/CIRCINTERVENTIONS.120.010296. Epub 2021 Oct 19. PMID 34665658
- [Background] Sato T, Yamamoto K, Matsumura M, Shlofmitz E, Khalique OK, Mintz GS, Shlofmitz RA, Jeremias A, Ali ZA, Maehara A. Discrimination of Calcified Nodule as a Cause of Coronary Angiographic Radiolucent Mass. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1948-1949. doi: 10.1016/j.jcin.2023.04.013. Epub 2023 Jul 5. No abstract available. PMID 37409997
- [Background] Sato T, Matsumura M, Yamamoto K, Shlofmitz E, Moses JW, Khalique OK, Thomas SV, Tsoulios A, Cohen DJ, Mintz GS, Shlofmitz RA, Jeremias A, Ali ZA, Maehara A. Impact of Eruptive vs Noneruptive Calcified Nodule Morphology on Acute and Long-Term Outcomes After Stenting. JACC Cardiovasc Interv. 2023 May 8;16(9):1024-1035. doi: 10.1016/j.jcin.2023.03.009. PMID 37164599
- [Background] Hada M, Kakuta T, Sugiyama T, Hoshino M, Yonetsu T, Usui E, Hanyu Y, Nagamine T, Nogami K, Ueno H, Matsuda K, Sayama K, Setoguchi M, Tahara T, Sakamoto T, Mineo T, Kobayashi N, Takano M, Kondo S, Wakabayashi K, Suwa S, Dohi T, Mori H, Kimura S, Mitomo S, Nakamura S, Higuma T, Yamaguchi J, Natsumeda M, Ikari Y, Yamashita J, Mizukami T, Yamamoto MH, Sasano T, Shinke T; TACTICS Investigators. Prognostic Impact of Culprit Lesion Calcified Nodule After Emergency Coronary Intervention: A TACTICS Registry Subanalysis. JACC Cardiovasc Imaging. 2024 Nov;17(11):1384-1386. doi: 10.1016/j.jcmg.2024.06.010. Epub 2024 Aug 7. No abstract available. PMID 39115502
- [Background] Madhavan MV, Alsaloum M, Maehara A, Gogia S, Lee J, Fall K, Prasad M, McEntegart MB, Kirtane AJ. Recurrent Calcified Nodule Protrusion Through Stent Struts After Percutaneous Coronary Intervention of the RCA. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2463-2465. doi: 10.1016/j.jcin.2023.07.033. Epub 2023 Sep 6. No abstract available. PMID 37676224
- [Background] Brott BC. The Calcified Nodule Paradox. JACC Cardiovasc Interv. 2023 May 8;16(9):1036-1038. doi: 10.1016/j.jcin.2023.04.001. No abstract available. PMID 37164600
- [Background] Shin D, Karimi Galougahi K, Spratt JC, Maehara A, Collet C, Barbato E, Ribichini FL, Gonzalo N, Sakai K, Mintz GS, Stone GW, Shlofmitz E, Shlofmitz RA, Jeremias A, Ali ZA. Calcified Nodule in Percutaneous Coronary Intervention: Therapeutic Challenges. JACC Cardiovasc Interv. 2024 May 27;17(10):1187-1199. doi: 10.1016/j.jcin.2024.03.032. PMID 38811101

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT07262359/Prot_SAP_ICF_000.pdf